CLINICAL TRIAL: NCT03685448
Title: A Phase II of Single Agent Cabozantinib in Patients With Locally Advanced or Metastatic Non-clear Cell Renal Cell Carcinoma Post Immunotherapy or Who Are Unsuitable for Immunotherapy (ANZUP1802)
Brief Title: ANZUP - Non-clear Cell Post Immunotherapy CABozantinib (UNICAB)
Acronym: UNICAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP1802
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma; Papillary Renal Cell Carcinoma Type 1; Papillary Renal Cell Carcinoma Type 2; Chromophobe Renal Cell Carcinoma; Sarcomatoid Renal Cell Carcinoma; Xp11.2 Translocation-Related Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Cabozantonib (Experimental): Cabozantinib 60 mg/day for up to 12 cycles (one cycle is 28 days), taken orally
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — The 20 mg cabozantinib drug product is a film-coated, white, round, immediate-release tablet. Cabozantinib should not be stored above 25°C (77°F).
  Other Names: Cabometyx

SUMMARY:
Renal cell carcinoma (RCC) is the 9th most common cancer in Australia, the 10th most common cancer in Western populations.~75% of kidney cancers are clear-cell renal cell carcinomas (ccRCC). Many patients present with advanced or unresectable disease at diagnosis and a number of treatments are now available for metastatic ccRCC included vascular endothelial growth factor receptor tyrosine kinase inhibitors (VEGFR TKIs), mTOR inhibitors, and cytokines. More recently first line use of immunotherapy demonstrated improved survival with checkpoint inhibitors. While many patients benefit from first-line treatment, progression is inevitable and these treatments remain on the whole palliative. Second-line VEGFR TKIs, mTOR inhibitors and immunotherapy have some benefit but in a smaller increment than first-line treatment.

While ~75% of kidney cancers are the clear-cell variant, ~25% of kidney cancers are non-clear cell histology (nccRCC) and include papillary, chromophobe, sarcomatoid, collecting duct carcinoma, Xp11 translocation carcinoma and unclassified. Patients with non-ccRCC have significantly lower response rates and poorer median progression-free survival and overall survival than those with ccRCC. Non clear cell histologies have largely been excluded from large phase III randomised clinical trials and therefore the optimal treatment and sequencing of therapies for these patients remains unclear.

Despite recent unprecedented advances in treatment, there continues to be an unmet need to improve outcomes for patients with previously untreated, unresectable or metastatic renal cell carcinoma. This is particularly relevant in non-clear cell RCC. Because it is a rarer subtype of metastatic renal cell carcinoma, it is more challenging to study, and treatment efficacy data is sparse.

The research project is testing a new treatment for participants with locally advanced or metastatic non-clear cell kidney cancer. The new treatment involves a drug called Cabozantinib (also known as Cabometyx). This drug has been used previously in many cancers, including clear cell kidney cancer and thyroid cancer.

The purpose of this study is to test the effectiveness (how well the drug works), safety, and tolerability of Cabozantinib. Cabozantinib is a anti-cancer drug that works by blocking cancer cell growth. It blocks particular proteins called protein kinases on cancer cells. Protein kinases encourage the cancer to grow. Cabozantinib is called a multi kinase inhibitor because it blocks a number of these proteins. How well cabozantinib works in cancer of the kidney will be tested by measuring the change in size of your tumours that are seen on CT scans.

Cabozantinib is approved to treat clear cell kidney cancer and thyroid cancer in Australia. It has not been tested in people with non-clear cell kidney cancer.

About 48 participants with non-clear cell kidney cancer are expected to participate in this study, from Australia. Even though this study may be suitable for you, it is possible that you may not be enrolled in this study.

This research study has been initiated by Dr. David Pook, is being conducted in collaboration with the Centre for Biostatistics and Clinical Trials (BaCT) and sponsored in Australia by the Australian and New Zealand Urogenital and Prostate (ANZUP) Cancer Trials Group Pty Ltd. Ipsen is supplying

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed un-resectable, locally advanced (defined as disease not amenable to curative surgery or radiation therapy) or metastatic non-clear cell renal cell histology (comprising greater than 50% of the tumour) including:

  1. Papillary renal cell carcinoma (type 1)
  2. Papillary renal cell carcinoma (type 2)
  3. Other subtypes: including chromophobe renal cell carcinoma, sarcomatoid renal cell carcinoma, Xp11 translocation (TFE3+ IHC) carcinoma, other renal carcinoma NOS
* Patient is either;

  1. Ineligible for checkpoint inhibitor immunotherapy due to pre-existing autoimmune disorder in the opinion of the investigator, or
  2. Has progressed following treatment with checkpoint inhibitor immunotherapy
* Be greater than 18 years of age on the day of signing informed consent
* At least 1 target lesion according to RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (refer to Appendix 1)
* Adequate bone marrow function (performed within 14 days prior to registration and with values within the ranges specified below):

  1. Haemoglobin ≥ 90g/L
  2. Platelets ≥ 100x109/L
  3. Neutrophil count ≥ 1.5x109/L
* Adequate liver function (performed within 14 days prior to registration and with values within the ranges specified below):

  1. Bilirubin ≤ 1.5 x upper limit of normal (ULN) except for participants with known Gilbert's syndrome who can have total bilirubin < 3.0 mg/dL
  2. AST or ALT ≤ 3.0 x ULN (or ≤ 5.0x ULN in the presence of liver metastases)
* Adequate renal function (performed within 14 days prior to registration and with values within the ranges specified below):

  1. Creatinine ≤ 1.5x ULN, or Creatinine clearance (CrCl) ≥ 30mL/min (use Cockcroft-Gault Formula, refer to Appendix 2)
  2. Urinalysis (dipstick) negative for protein, or for those with positive protein detected on urinalysis (≥2+), urine protein-to-creatinine ratio (UPCR) ≤ 1mg/mg (≤ 113.2mg/mmol)
* Negative pregnancy test for female participants of childbearing potential within 72 hours prior to registration. If urine test cannot be confirmed as negative, a negative serum pregnancy test is required.
* Female participants of childbearing potential must be willing to use two methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for greater than 1 year.
* Male participants with sexual partners of childbearing age must agree to use an adequate method of contraception, must agree to use a condom during intercourse and must agree to refrain from sperm donation starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Able to provide a formalin-fixed paraffin embedded (FFPE) tumour block, representative of the participant's primary or metastatic disease (preferred), which must be forwarded to the Centre for Biostatistics and Clinical Trials (BaCT) within 10 working days post registration (if not previously collected for the UNISoN study). Note: If FFPE tumour tissue block is not obtainable, then unstained slides are also acceptable. If archival tissue is not available, patient must be willing to provide a fresh tumour biopsy.
* Willing and able to start treatment within 14 days of registration, and to comply with all study requirements, including the timing and/or nature of the required treatment and assessments
* Has provided signed, written informed consent.

Exclusion Criteria:

* Patients with urothelial or transitional cell carcinoma of the renal pelvis or ureter
* Predominant clear cell renal cell carcinoma. A minority of clear cell histology (<50%) is acceptable, but there must be >50% non-clear cell histology predominant.
* Untreated brain or leptomeningeal metastases or current clinical or radiological progression of known brain metastases or requirement for steroid therapy for brain metastases. Participants with treated brain metastases are eligible if metastases have been shown to be stable on repeat imaging post treatment and steroid treatment has been ceased for ≥ 3 weeks.
* Serious Cardiovascular disorders:

  1. Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
  2. Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
  3. Stroke (including TIA), myocardial infarction, or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before randomization.
* Active infection requiring systemic therapy within 14 days before registration.
* Concurrent treatment with strong CYP3A4 inducers or inhibitors (such as ketoconazole and rifampicin), P-glycoprotein substrates (such as fexofenadine, ambrisentan, dabigatran etexilate, digoxin, colchicine, maraviroc, posaconazole, ranolazine, saxagliptin, sitagliptin, talinolol and tolvaptan), MRP2 inhibitors (such as cyclosporine, efavirenz and emtricitabine), or direct oral anticoagulants such as thrombin inhibitors or factor Xa inhibitors. Use of low molecular weight heparin (LMWH) is permitted.
* Life expectancy of less than 3 months.
* Prior systemic therapy, surgery or radiation therapy within 4 weeks before registation. Note: If the participant has undergone major surgery, complete wound healing must have occurred 1 month prior to registration. Patients must not have received prior targeted therapy or chemotherapy, but may have received previous checkpoint immunotherapy, for example, via the UNISoN trial (NCT03177239)
* History of another active malignancy except for locally curable cancers that have been apparently cured, such as low-grade thyroid carcinoma, prostate cancer not requiring treatment (Gleason grade ≤ 6), basal or squamous cell skin cancer, superficial bladder cancer, melanoma in situ or carcinoma in situ of the prostate, cervix, or breast. Participants who have been treated for other malignancies and have a <5% chance of relapse according to the investigator are eligible for this study.
* Other significant active infection, including hepatitis B, hepatitis C and HIV. Hepatitis and HIV testing is not mandatory unless clinically indicated.
* Participants should be excluded if they have a history of allergy to study drug components or problems of galactose intolerance, the Lapp lactase deficiency or glucose galactose malabsorption
* Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol
* Patient is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
The objective response rate (ORR), as assessed by RECIST 1.1. | Through study completion, on average 2 years.
  This is defined as the proportion of participants in the analysis set with a confirmed complete response (CR) or partial response (PR) divided by the number of participants in the analysis set.

SECONDARY OUTCOMES:
The number of participants with adverse events that are related to study drug, as assessed and graded by CTCAE v5.0. | From time of patient registration, until 30 days after the last dose of treatment.
Progression-free survival (PFS), as assessed by RECIST1.1. | Through study completion, on average 2 years.
The number of patients alive at the end of the study, as assessed by date of death. Overall survival (OS) is defined as the time between the date of registration to part 1 of the study and the date of death due to any cause. | Through study completion, on average 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: David Pook, MBBS FRACPMD, Principal Investigator — Australian & New Zealand Urogenital & Prostate Cancer Trials Group
Locations (11):
- Australia (11):
  - Border Medical Oncology Research Unit / The Border Cancer Hospital, Albury, New South Wales
  - Campbelltown Hospital, Campbelltown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Adelaide Cancer Centre / Ashford Cancer Centre Research / Cancer Care SA, Kurralta Park, South Australia
  - Box Hill Hospital - Eastern Health, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Goulburn Valley Health, as a satellite site under the supervision of Border Medical Oncology Research Unit, via the Tele-trial model, Shepparton, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — https://anzup.org.au/